CLINICAL TRIAL: NCT02232100
Title: Internet-Delivered Attentional Bias Modification Training in People With Chronic Musculoskeletal Pain: A Double-Blind Randomised Control Trial and a Qualitative Investigation of Participants' Experience.
Brief Title: Attentional Bias Modification Training for People With Chronic Musculoskeletal Pain
Acronym: I-ABMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABMT2014
Record Dates: First submitted 2014-09-01; First posted 2014-09-04 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Chronic Pain
Keywords: Attentional bias modification training; Chronic pain; Visual-probe task; Internet-delivered therapy
MeSH Terms: conditions — Chronic Pain | interventions — acceleratory factor from growth hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 10AMG (Experimental): Attentional bias modification group - 10 training sessions
  Interventions: Behavioral: Attentional bias modification training (AMG)
- 10ACG (Placebo Comparator): Attentional control group - 10 placebo sessions
  Interventions: Behavioral: Attentional bias placebo (ACG)
- 18AMG (Experimental): Attentional bias modification group - 18 training sessions
  Interventions: Behavioral: Attentional bias modification training (AMG)
- 18ACG (Placebo Comparator): Attentional control group - 18 placebo sessions
  Interventions: Behavioral: Attentional bias placebo (ACG)

INTERVENTIONS:
Behavioral: Attentional bias modification training (AMG) — Attentional bias modification, administered via an internet-delivered visual-probe task that trains attention away from pain-related information
  Arms: 10AMG; 18AMG
Behavioral: Attentional bias placebo (ACG) — Attentional bias placebo, administered via an internet-delivered visual-probe task that does not train attention either away or towards pain-related information
  Arms: 10ACG; 18ACG

SUMMARY:
Chronic musculoskeletal pain is a complex medical condition associated with significant distress, disability, and reduction in quality of life. Research has shown that patients with chronic musculoskeletal pain demonstrate attentional biases towards pain-related information.

The purpose of this study is to determine whether internet-delivered attentional bias modification, which aims to implicitly train attention away from pain-related information, has beneficial effects upon pain and pain-related distress in patients with chronic musculoskeletal pain.

Participants will be randomised to either an attentional training condition, or to a no-training placebo condition. The primary outcome measures are pain intensity and pain interference, and secondary outcome measures include anxiety, depression, pain-related fear and sleep problems.

Data will be analysed and reported separately for participants aged 16 - 24 and 25 - 60. It is hypothesized that participants receiving internet-delivered attentional bias modification will show significantly greater reductions in pain and pain-related distress compared to participants receiving placebo training.

DETAILED DESCRIPTION:
Chronic musculoskeletal pain is a complex medical condition. Patients often experience increased levels of pain-related distress, including anxiety, depression and disability, impaired sleep, poor well-being and diminished quality of life. Over the past decade, numerous studies have provided evidence for the existence of attentional bias towards pain-related information in chronic pain patients. A critical question remaining unanswered is whether pain-related bias is simply an epiphenomenon of chronic pain, or whether it has a causal role in the maintenance of pain. Recently, there has been growing interest in the potential benefits of attentional retraining in individuals with various emotional disorders, with focus upon attentional bias modification (ABM).

ABM is a theory-driven intervention which uses computer-based paradigms, typically the visual-probe task, to implicitly manipulate attention away from sources of threat relevant to the individual's fears or concerns. To date, three published studies using ABM with chronic pain patients exist, the combined results of which support the therapeutic benefits of ABM on pain, pain-related distress and disability. Considering these encouraging results, it is important to expand this field of research and explore ABM in chronic pain in greater depth. In particular, all former studies assessed the clinical effectiveness of ABM in laboratory environments. The purpose of this double-blind RCT study is to determine whether internet-delivered ABM training (I-ABMT) has therapeutic benefits for patients with chronic musculoskeletal pain on pain and pain-related distress, thereby assessing training effects in real-world settings.

The visual-probe task will be used for assessment and modification of pain-related attentional biases. This is a computerised paradigm which records participant response times to a series of visual stimuli. Following an initial fixation point, each trial presents a stimulus pair in distinct locations (e.g. left and right of the initial fixation point), for a specified length of time (i.e., 500 or 1250ms). Stimuli may consist of words or images, with experimental trials featuring one pain-related stimulus and one neutral stimulus. Following this, both stimuli are removed, with a visual probe replacing one stimulus. Participants indicate the location of this probe as quickly and accurately as possible via manual response. Response times are faster to probes appearing in an attended region of the screen than an unattended region, providing a measure of attentional allocation. Averaged response times are calculated, which are converted into an index of attentional bias. In the standard and control (i.e., placebo) versions of the visual probe task, the probe replaces pain-related and neutral stimuli an equal number of times, while in the I-ABMT version, the probe always replaces neutral stimuli thus training attention away from pain-related stimuli.

Dose effects will be explored in this study, with participants randomised to one of four conditions: (i) 10-session Attentional Modification Group , (ii) 10-session Attentional Control Group, (iii) 18-session Attentional Modification Group, and (iv) 18-session Attentional Control Group. The primary outcome measures are pain intensity and pain interference, and secondary outcome measures include anxiety, depression, pain-related fear and sleeping impairment, including engagement to and satisfaction with the online visual-probe training task. It is hypothesized that participants receiving ABM training will show significantly greater reductions in pain and pain-related distress compared to participants receiving placebo training. Dose effects will be investigated in an exploratory manner, and data will be analysed and reported separately for participants aged 16 - 24 and 25 - 60.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 16 to 60 years old
2. experiencing any type of CMSK (i.e., any condition that involves pain lasting for more than three months and arises from bones, muscles and/or joints)
3. able to sit at a personal computer for forty minutes
4. normal or corrected to normal vision
5. access to the internet at least twice a week
6. access to, and familiarity using, a Windows-based computer (g) successful completion of primary school
7. living in the United Kingdom.

Exclusion Criteria:

1. experiencing malignant CMSK (i.e., pain caused due to a tumour)
2. a diagnosis of any psychiatric disorder, either currently or within the last 5 years
3. currently under psychiatric therapy.

No restrictions are placed on concomitant care and participants are not required to make any changes to current treatments they may be receiving.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity - change from baseline on an 11-point scale (0 no pain, 10 pain as bad as you can imagine) to endline (4 or 8 weeks) | Baseline, following intervention (4 or 8 weeks)
  Likert scale from the Brief Pain Inventory-Short Form (BPS-SF), a commonly used measure of pain intensity and pain interference.
Pain interference- change from baseline on an 11-point scale (0 does not interfere, 10 completely interferes) to endline (4 or 8 weeks) | Baseline, following intervention (4 or 8 weeks)
  Likert scale from the Brief Pain Inventory-Short Form (BPS-SF), a commonly used measure of pain intensity and pain interference.
Pain intensity - change from baseline on an 11-point scale (0 no pain, 10 pain as bad as you can imagine) to 6-month follow-up | Baseline, 6-month follow-up
  Likert scale from the Brief Pain Inventory-Short Form (BPS-SF), a commonly used measure of pain intensity and pain interference.
Pain interference- change from baseline on an 11-point scale (0 does not interfere, 10 completely interferes) to 6-month follow-up | Baseline, 6-month follow-up
  Likert scale from the Brief Pain Inventory-Short Form (BPS-SF), a commonly used measure of pain intensity and pain interference.

SECONDARY OUTCOMES:
Anxiety - change from baseline to endline (4 or 8 weeks) | Baseline, following intervention (4 or 8 weeks)
  State and Trait Anxiety Subscales from the State-Trait Anxiety Inventory (STAI), a 40-item measure of state and trait anxiety (20 items each). Each item is measured on a four point scale, with possible scores for both state and trait levels ranging between 20 and 80. State and trait subscales are not combined. Higher scores on each subscale represent more intense or more frequent feelings of anxiety.
Depression - change from baseline to endline (4 or 8 weeks) | Baseline, following intervention (4 or 8 weeks)
  Depression Subscale from Hospital Anxiety and Depression Scale, which is comprised of 7 items each measured on a four point scale. Possible scores for the depression subscale range between 0 and 21, with higher scores indicating higher levels of anxiety and depression.
Pain-related fear - change from baseline to endline (4 or 8 weeks) | Baseline, following intervention (4 or 8 weeks)
  Fear of Pain questionnaire III. On a 5-point scale, respondents are asked to rate how fearful they are of pain associated with specific situations and events (e.g., being in an automobile accident). Possible scores range between 30 and 150, with higher scores representing a more intense fear of pain. In addition to a total score, the measure also provides subscales of minor, severe, and medical pain-related fear.
Sleeping impairment - change from baseline to endline (4 or 8 weeks) | Baseline, following intervention (4 or 8 weeks)
  Medical Outcome Study Sleep Scale, a twelve-item questionnaire developed for patients with chronic illness, measuring six dimensions of sleep over the past four weeks; sleep initiation (time to fall asleep - five responses), quantity (the participant writes hours per night sleeping), maintenance, respiratory problems, perceived adequacy, and somnolence rated on a 6-point scale. A sleep problems index which summarises information from nine items is also be scored. Responses are recoded on a 0 - 100 scale, with higher scores indicating more of the concept being measured (e.g., greater difficulties falling asleep).
Anxiety - change from baseline to 6-month follow-up | Baseline, 6-month follow-up
  State and Trait Anxiety Subscales from State-Trait Anxiety Inventory(STAI), a 40-item measure of state and trait anxiety (20 items each). Each item is measured on a four point scale, with possible scores for both state and trait levels ranging between 20 and 80. State and trait subscales are not combined. Higher scores on each subscale represent more intense or more frequent feelings of anxiety.
Depression - change from baseline to 6-month follow-up | Baseline, 6-month follow-up
  Depression Subscale from Hospital Anxiety and Depression Scale, which is comprised of 7 items each measured on a four point scale. Possible scores for the depression subscale range between 0 and 21, with higher scores indicating higher levels of anxiety and depression.
Pain-related fear - change from baseline to 6-month follow-up | Baseline, 6-month follow-up
  Fear of Pain questionnaire III. On a 5-point scale, respondents are asked to rate how fearful they are of pain associated with specific situations and events (e.g., being in an automobile accident). Possible scores range between 30 and 150, with higher scores representing a more intense fear of pain. In addition to a total score, the measure also provides subscales of minor, severe, and medical pain-related fear.
Sleeping impairment - change from baseline to 6-month follow-up | Baseline, 6-month follow-up
  Medical Outcome Study Sleep Scale, a twelve-item questionnaire developed for patients with chronic illness, measuring six dimensions of sleep over the past four weeks; sleep initiation (time to fall asleep - five responses), quantity (the participant writes hours per night sleeping), maintenance, respiratory problems, perceived adequacy, and somnolence rated on a 6-point scale. A sleep problems index which summarises information from nine items is also be scored. Responses are recoded on a 0 - 100 scale, with higher scores indicating more of the concept being measured (e.g., greater difficulties falling asleep).

OTHER OUTCOMES:
Satisfaction with the online ABMT | Following intervention (4 or 8 weeks)
  Satisfaction with the online treatment questionnaire. Participants state how strongly they agree/disagree with each of the following items: (a) the use of a computer to access treatment, (b) level of easiness of the online intervention, (c) duration of the potential effects of the treatment, and (d) potential recommendation of online interventions to others. Responses are provided on a 5-point scale ranging from "Agree very strongly" to "Disagree very strongly". An additional question asks participants how helpful they have found the online intervention, with responses provided on a 4-point scale ranging from "Very helpful" to "Not at all helpful". Two open questions are also included that require participants to state the aspects of the intervention they most liked and disliked.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Liossi, DPsych, Principal Investigator — University of Southampton
Locations (1):
- University of Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liossi C, Georgallis T, Zhang J, Hamilton F, White P, Schoth DE. Internet-delivered attentional bias modification training (iABMT) for the management of chronic musculoskeletal pain: a protocol for a randomised controlled trial. BMJ Open. 2020 Feb 20;10(2):e030607. doi: 10.1136/bmjopen-2019-030607. PMID 32086350